CLINICAL TRIAL: NCT04466891
Title: A Phase 2b, Open-label, Single-arm Study of ZW25 Monotherapy in Subjects With Advanced or Metastatic HER2-amplified Biliary Tract Cancers
Brief Title: A Study of ZW25 (Zanidatamab) in Subjects With Advanced or Metastatic HER2-Amplified Biliary Tract Cancers
Acronym: HERIZON-BTC-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: BeiGene (Industry); Jazz Pharmaceuticals Ireland Limited (Industry); BeOne Medicines LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW25-203; 2020-000459-11 (EudraCT Number)
Expanded Access: NCT04578444 (No longer available)
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: HER2-amplified Biliary Tract Cancers
Keywords: HER2; Bispecific antibody; Biparatopic antibody; Immunotherapy; Biliary Tract Cancer; Intra-hepatic cholangiocarcinoma; Extra-hepatic cholangiocarcinoma; Gallbladder cancer; JZP598
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms | interventions — zanidatamab

STUDY DESIGN:
Intervention Model Description: single-arm, open-label, multi-cohort, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZW25 (Zanidatamab) Monotherapy (Experimental)
  Interventions: Drug: ZW25 (Zanidatamab)

INTERVENTIONS:
Drug: ZW25 (Zanidatamab) — Administered intravenously
  Other Names: JZP598; ZW25; ZIIHERA®

SUMMARY:
This multicenter, open-label, single-arm trial will evaluate the anti-tumor activity of ZW25 (zanidatamab) monotherapy in subjects with human epidermal growth factor receptor 2 (HER2)-amplified, inoperable and advanced or metastatic biliary tract cancer (BTC), including intra-hepatic cholangiocarcinoma (ICC), extra-hepatic cholangiocarcinoma (ECC), and gallbladder cancer (GBC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed BTC, including ICC, ECC or GBC.
* Locally advanced or metastatic BTC and not eligible for curative resection, transplantation, or ablative therapies.
* Received at least 1 prior gemcitabine-containing systemic chemotherapy regimen for advanced disease, and experienced disease progression after or developed intolerance to the most recent prior therapy. For subjects who received gemcitabine in prior adjuvant or neoadjuvant treatment, if progression occurred < 6 months from the latter of primary surgical resection or completion of gemcitabine-containing adjuvant therapy, they will be considered as having received 1 prior line of therapy for advanced disease.
* Subjects must test positive for HER2 amplification by ISH-assay at a central laboratory on a new biopsy or archival tissue. Note that fine needle aspirates (FNAs; cytology samples) and biopsies from sites of bone metastases are not acceptable. Testing may occur at any time after diagnosis of advanced or metastatic disease and before study enrollment.
* Male or female, ≥18 years of age (or the legal age of adulthood per country-specific regulations).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Adequate organ function.
* Adequate cardiac function, as defined by left ventricular ejection fraction ≥ 50%.

Exclusion Criteria:

* Received systemic anti-cancer therapy within 3 weeks of the first dose of ZW25. Received radiotherapy within 2 weeks of the first dose of ZW25.
* Prior treatment with HER2-targeted agents.
* Untreated central nervous system (CNS) metastases, symptomatic CNS metastases, or radiation treatment for CNS metastases within 4 weeks of start of study treatment. Stable, treated brain metastases are allowed (defined as subjects who are off steroids and anticonvulsants and are neurologically stable with no evidence of radiographic progression for at least 4 weeks at the time of screening).
* Known leptomeningeal disease (LMD). If LMD has been reported radiographically on baseline MRI, but is not suspected clinically by the investigator, the subject must be free of neurological symptoms of LMD.
* Concurrent uncontrolled or active hepatobiliary disorders or untreated or ongoing complications after laparoscopic procedures or stent placement, including but not limited to active cholangitis, unresolved biliary obstruction, infected biloma or abscess. Any complications must be resolved more than 2 weeks prior to the first dose of ZW25.
* Prior or concurrent malignancy whose natural history or treatment has, in the opinion of the investigator or medical monitor, the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Active hepatitis
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2
* QTc Fridericia (QTcF) > 470 ms.
* History of myocardial infarction or unstable angina within 6 months prior to enrollment, troponin levels consistent with myocardial infarction, or clinically significant cardiac disease.
* Acute or chronic uncontrolled pancreatitis or Child-Pugh Class C liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (14):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Advent Health Cancer Institute, Orlando, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center - Hospital, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Chile (2):
  - Centro de Cáncer Nuestra Señora de la Esperanza, Santiago
  - Radiomed (Clinica Alemana de Temuco), Temuco
- China (23):
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Chengdu
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Hospital, Hefei
  - Huzhou Central Hospital, Huzhou
  - Jinhua Central Hospital, Jinhua
  - The First Hospital Of Lanzhou University, Lanzhou
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Shandong Provincial Third Hospital, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai
  - The Third Affiliated Hospital of the Chinese PLA, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- France (5):
  - Oncologie médicale Hopital Jean Minjoz, Besançon
  - Institut de Cancerologie et d'Hematologie Hopital Morvan - CHRU de Brest, Brest
  - Hopitaux de La Timone, Marseille
  - Département Oncologie Gastro-entérologie CHRU de Poitiers La Miletrie, Poitiers
  - Département De Médecine, Villejuif
- Italy (4):
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo
  - Istituto Clinico Humanitas, Milan
  - Istituto Nazionale Dei Tumori, Milan
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua
- South Korea (8):
  - Gyeongsang National University Hospital, Jinju
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (3):
  - University College London Hospitals (UCLH), London
  - Royal Free London NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing

REFERENCES:
- [Derived] Harding JJ, Fan J, Oh DY, Choi HJ, Kim JW, Chang HM, Bao L, Sun HC, Macarulla T, Xie F, Metges JP, Ying J, Bridgewater J, Lee MA, Tejani MA, Chen EY, Kim DU, Wasan H, Ducreux M, Bao Y, Lindsey S, Bachini M, Morement H, Boyken L, Ma J, Garfin P, Pant S; HERIZON-BTC-01 study group. A plain language summary of the results from the phase 2b HERIZON-BTC-01 study of zanidatamab in participants with HER2-amplified biliary tract cancer. Future Oncol. 2024;20(31):2319-2329. doi: 10.1080/14796694.2024.2368952. Epub 2024 Aug 8. PMID 39114870
- [Derived] Harding JJ, Fan J, Oh DY, Choi HJ, Kim JW, Chang HM, Bao L, Sun HC, Macarulla T, Xie F, Metges JP, Ying J, Bridgewater J, Lee MA, Tejani MA, Chen EY, Kim DU, Wasan H, Ducreux M, Bao Y, Boyken L, Ma J, Garfin P, Pant S; HERIZON-BTC-01 study group. Zanidatamab for HER2-amplified, unresectable, locally advanced or metastatic biliary tract cancer (HERIZON-BTC-01): a multicentre, single-arm, phase 2b study. Lancet Oncol. 2023 Jul;24(7):772-782. doi: 10.1016/S1470-2045(23)00242-5. Epub 2023 Jun 2. PMID 37276871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 87 participants who met all eligibility criteria were enrolled and received treatment.
Pre-assignment Details: Participants must have received at least 1 prior gemcitabine-containing systemic chemotherapy regimen for advanced disease and experienced disease progression after or developed intolerance to the most recent prior therapy.
Groups:
- Cohort I: Participants with advanced or metastatic biliary tract cancer with HER2 amplification by in situ hybridization (ISH) and HER2 overexpression by immunohistochemistry (IHC) which includes IHC 2+ or 3+
- Cohort II: Participants with advanced or metastatic biliary tract cancer with HER2 amplification by ISH and HER2 IHC 0 or 1+.
Period: Overall Study
Arm/Group | Cohort I | Cohort II
Started | 80 | 7
Completed | 0 | 0
Not Completed | 80 | 7
Not completed — Death | 60 | 6
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Study terminated by sponsor | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Transitioned to Named Patient Supply (NPS) program | 5 | 0

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I | Cohort II | Total
Number analyzed (Participants) | 80 | 7 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.56) | 65.4 (8.75) | 62.7 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 2 | 47
  Male | 35 | 5 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 72 | 6 | 78
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 52 | 5 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 2 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) by Independent Central Review (ICR)
Description: Number of participants who achieved a confirmed best overall response (BOR) of either complete response (CR) or partial response (PR) during treatment per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response (CR) is defined as a disappearance of all target and non-target lesions and partial response (PR) is defined as at least a 30% decrease in the sum of diameters of all target lesions.
Time Frame: Up to 34 months
Population: Assessed in participants with available data in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
Participants | 33 | 0

2. Secondary Outcome: Duration of Response (DOR) by ICR
Description: The time from the first confirmed objective response (CR or PR) to documented progressive disease (PD) per RECIST 1.1, or death from any cause
Time Frame: Up to 45 months
Population: Only participants with a response (a confirmed Complete Response (CR) or confirmed Partial Response (PR)), as evaluated by ICR, were evaluated for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 33 | 0
months | 14.92 [7.39 to 23.98] |

3. Secondary Outcome: DOR ≥ 16 Weeks by ICR
Description: Proportion of subjects with a DOR ≥ 16 weeks per RECIST 1.1
Time Frame: 24 weeks, up to 45 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 33 | 0
Participants | 28 |

4. Secondary Outcome: Disease Control Rate (DCR) by ICR
Description: Number of subjects who achieved a best overall response of stable disease (SD), non-CR/non-PD, or confirmed CR or PR per RECIST 1.1
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
Participants | 55 | 3

5. Secondary Outcome: Progression-free Survival (PFS) by ICR
Description: The time from the first dose of study treatment to the date of documented disease progression (per RECIST 1.1), or death from any cause
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
months | 5.49 [3.65 to 7.29] | 1.87 [1.22 to NA] — Upper Confidence Interval (CI) not estimable due to insufficient events

6. Secondary Outcome: ORR by Investigator Assessment
Description: Number of subjects who achieved a confirmed BOR of either CR or PR during treatment per RECIST 1.1
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
Participants | 34 | 0

7. Secondary Outcome: DOR by Investigator Assessment
Description: as for outcome 2
Time Frame: Up to 45 months
Population: Only participants with a response (a confirmed Complete Response (CR) or confirmed Partial Response (PR)) as per investigator assessment, were evaluated for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 34 | 0
months | 11.10 [7.46 to 14.06] |

8. Secondary Outcome: DOR ≥ 16 Weeks by Investigator Assessment
Description: Proportion of subjects with a DOR ≥ 16 weeks per RECIST 1.1
Time Frame: 24 weeks, up to 45 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 34 | 0
Participants | 31 |

9. Secondary Outcome: DCR by Investigator Assessment
Description: as for outcome 4
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
Participants | 54 | 1

10. Secondary Outcome: PFS by Investigator Assessment
Description: as for outcome 5
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
months | 5.37 [3.55 to 7.29] | 1.77 [0.79 to 1.94]

11. Secondary Outcome: Overall Survival
Description: The time from the first dose of study treatment until the date of death from any cause
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
months | 15.54 [10.38 to 18.66] | 5.52 [1.22 to NA] — Upper CI not estimable due to insufficient events

12. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Number of subjects who experienced AEs or serious adverse events
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
Participants
  Any Treatment Emergent Adverse Event (TEAE) | 78 | 6
  Zanidatamab related TEAE | 61 | 2
  Any Treatment Emergent Serious Adverse Event | 43 | 3
  Zanidatamab related serious TEAE | 8 | 0
  Zanidatamab related TEAE resulting in treatment discontinuation | 2 | 0

13. Secondary Outcome: Incidence of Laboratory Abnormalities
Description: Number of subjects who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
Participants | 37 | 7

14. Secondary Outcome: Maximum Serum Concentration of ZW25
Time Frame: Pre-dose, end of infusion, 2, 4, 8, 24 and 96 hours post dose
Population: All subjects who received any amount of zanidatamab and have at least 1 post-baseline PK assessment were included in this outcome
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
micrograms per milliliter | 457.6 (15.44) | 443.6 (24.10)

15. Secondary Outcome: Trough Concentration of ZW25
Description: Minimum observed serum concentration (trough)
Time Frame: Pre-dose, end of infusion, 2, 4, 8, 24 and 96 hours post dose
Population: All subjects who received any amount of zanidatamab and have at least 1 post-baseline pharmacokinetic (PK) assessment were included in this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 80 | 7
micrograms per milliliter | 73.4 (42.10) | 46.5 (18.66)

16. Secondary Outcome: Incidence of Anti-drug Antibodies (ADAs)
Description: Number of subjects who develop ADAs
Time Frame: Up to 45 months
Population: All subjects who received any amount of zanidatamab and have both baseline anti-drug antibodies (ADA) and at least 1 post baseline ADA results available were included in this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 78 | 7
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of dosing of any study drug up until 30 days after last study dose, up to approximately 45 months
Arm/Group | Cohort I | Cohort II
All-Cause Mortality (participants affected / at risk) | 60/80 | 6/7
Serious Adverse Events (participants affected / at risk) | 43/80 | 3/7
Other Adverse Events (participants affected / at risk) | 78/80 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (N=80) | Cohort II (N=7)
Jaundice cholestatic (Hepatobiliary disorders) | 5 | 0
Biliary obstruction (Hepatobiliary disorders) | 4 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 2
Jaundice (Hepatobiliary disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 4 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Biliary sepsis (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Cholangitis infective (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Haematochezia (Hepatobiliary disorders) | 1 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (N=80) | Cohort II (N=7)
Anemia (Blood and lymphatic system disorders) | 18 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 16 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0
Ascites (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 39 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 14 | 0
Vomiting (Gastrointestinal disorders) | 13 | 1
Asthenia (General disorders) | 6 | 1
Fatigue (General disorders) | 11 | 0
Oedema peripheral (General disorders) | 5 | 0
Pyrexia (General disorders) | 14 | 0
Drug hypersensitivity (Immune system disorders) | 3 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 27 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 16 | 1
Aspartate aminotransferase increased (Investigations) | 15 | 1
Blood alkaline phosphatase increased (Investigations) | 7 | 2
Blood bilirubin increased (Investigations) | 10 | 0
Blood creatinine increased (Investigations) | 6 | 1
Ejection fraction decreased (Investigations) | 11 | 0
Gamma-glutamyltransferase increased (Investigations) | 6 | 1
Neutrophil count increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 11 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 11 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1
Hypoproteinemia (Metabolism and nutrition disorders) | 1 | 1
Dizziness (Nervous system disorders) | 7 | 0
Peripheral sesory neuropathy (Nervous system disorders) | 6 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 11 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 0
Hypertension (Vascular disorders) | 10 | 0
COVID-19 (Infections and infestations) | 5 | 1
Insomnia (Psychiatric disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT04466891/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04466891/SAP_001.pdf